CLINICAL TRIAL: NCT02701725
Title: Compensatory Reserve Index as a Hemodynamic Status Evaluation Tool in Patients
Acronym: CRIHEM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0260-15-MMC
Record Dates: First submitted 2016-03-01; First posted 2016-03-08 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Hemorrhage; Sepsis
MeSH Terms: conditions — Hemorrhage; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CRI status — Measurement of CRI

SUMMARY:
The investigators will use the Compensatory Reserve Index (CRI) device to monitor hemodynamic status of patients in the hospital. CRI values of patients will be monitored during their care in order to verify the compliance of the values to the physiological condition. During the protocol investigators will document patients injuries, life-saving procedures performed, response to treatment as well progress to systemic inflammatory response syndrome (SIRS) and sepsis.

The indices measured in the study will not be a consideration when handling patients. The medical team will not be exposed to metrics measured.

DETAILED DESCRIPTION:
Assessment of patients in the emergency department, ICU or surgical department can be a challenging process. This assessment includes collecting data regarding injury mechanism, vital signs, and physical examination findings before proceeding to other ways of evaluating the patient.

These data are then integrated in an attempt to form an accurate patient status and to determine the urgency of treatment and evacuation to the next echelon of care when necessary. When caring for multiple casualties, this process takes on an even greater importance because the care of one patient can delay the care of others.

Triage and monitoring of patients consists of several vital sign measurements including blood pressure, oxygen saturation, and heart rate. These measurements show varying correlation with patient survival, Injury Severity Score, and the need for life-saving intervention. The most significant disadvantage of their use as part of patient triage is that they are all retrospective by nature, and a change in these indices occur only after substantial hemodynamic compromise and failure of compensatory mechanisms when life-saving interventions might be too late.

Because of the limitations inherent to these vital signs, several calculated indices have been suggested in an attempt to integrate a few vital signs into more sensitive metrics for prediction of patient outcomes. The most frequently described metric is shock index (SI), which is calculated as the ratio between heart rate and systolic blood pressure (normal values, 0.5 Y 0.7), and has demonstrated superiority over other indices. Heart rate variability has also been frequently suggested as a calculated vital sign, but its clinical utility in the acute blood loss setting has proven to be limited as a result of its high interpatient and intrapatient variability.

The Compensatory Reserve Index (CRI) represents a new paradigm for measuring the physiological reserve of integrated cardiopulmonary mechanisms (e.g., tachycardia, vasoconstriction, breathing) that compensate for reduced central blood volume. Advanced sensor technologies such as photoplethysmography enable noninvasive recordings of analog arterial waveforms. Using a model that induces stepwise reduction of central blood volume (lower body negative pressure [LBNP]) in volunteering young healthy human test subjects, through application of negative pressure to the lower body, feature-extraction and machine-learning techniques were used to reveal subtle changes in waveform features that are associated with a declining volume. This approach enables simultaneous abstraction and normalization of various characteristics of the arterial waveform. As such, the CRI aims to reflect the capacity of all factors contributing to physiological compensatory mechanisms, including compensatory reflexes, various muscle contractions, and respirations, among others. Compensatory Reserve Index values range from 0 (complete decompensation) to 1 (full compensatory reserve available). The device itself is compact, light, and can be placed on the patient's finger, and the test can be performed within 30 s, making the measurement of CRI theoretically feasible in almost any setting. The approach was designed to prospectively identify ongoing loss of central blood volume and thus estimate the point at which individuals will experience hemodynamic decompensation (onset of shock) well in advance compared with changes in standard or "legacy" vital signs.

The CRI has been shown to correlate with central blood volume changes in human subjects in laboratory conditions however, few published data regarding its use in other experimental models or its ability to detect actual blood loss exist. The current investigation represents the first effort to apply a small pulse oximeter unit to test the CRI on human subjects admitted to hospital.

The purpose of the study is to test the hypothesis that a novel noninvasive CRI monitoring algorithm would demonstrate greater sensitivity and specificity compared with standard vital signs for identifying patients with blood loss, SIRS, sepsis thus enabling appropriate measures to be taken.

ELIGIBILITY:
Inclusion Criteria:

* All patients with blood loss (trauma or disease)
* All patients receiving blood products of any type
* All patients with SIRS or Sepsis
* All patients who are anticipated to suffer for sepsis

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective Review of all adult patients admitted to Meir Medical Center who meet criteria.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-05 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
change in CRI | 6 m

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King DR, Ogilvie MP, Pereira BM, Chang Y, Manning RJ, Conner JA, Schulman CI, McKenney MG, Proctor KG. Heart rate variability as a triage tool in patients with trauma during prehospital helicopter transport. J Trauma. 2009 Sep;67(3):436-40. doi: 10.1097/TA.0b013e3181ad67de. PMID 19741382
- [Background] Convertino VA, Ryan KL, Rickards CA, Salinas J, McManus JG, Cooke WH, Holcomb JB. Physiological and medical monitoring for en route care of combat casualties. J Trauma. 2008 Apr;64(4 Suppl):S342-53. doi: 10.1097/TA.0b013e31816c82f4. PMID 18385586
- [Background] Soller BR, Zou F, Ryan KL, Rickards CA, Ward K, Convertino VA. Lightweight noninvasive trauma monitor for early indication of central hypovolemia and tissue acidosis: a review. J Trauma Acute Care Surg. 2012 Aug;73(2 Suppl 1):S106-11. doi: 10.1097/TA.0b013e318260a928. PMID 22847078
- [Background] Bruijns SR, Guly HR, Bouamra O, Lecky F, Lee WA. The value of traditional vital signs, shock index, and age-based markers in predicting trauma mortality. J Trauma Acute Care Surg. 2013 Jun;74(6):1432-7. doi: 10.1097/TA.0b013e31829246c7. PMID 23694869
- [Background] Moulton SL, Mulligan J, Grudic GZ, Convertino VA. Running on empty? The compensatory reserve index. J Trauma Acute Care Surg. 2013 Dec;75(6):1053-9. doi: 10.1097/TA.0b013e3182aa811a. PMID 24256681
- [Background] Birkhahn RH, Gaeta TJ, Terry D, Bove JJ, Tloczkowski J. Shock index in diagnosing early acute hypovolemia. Am J Emerg Med. 2005 May;23(3):323-6. doi: 10.1016/j.ajem.2005.02.029. PMID 15915406
- [Background] Rixen D, Siegel JH, Friedman HP. "Sepsis/SIRS," physiologic classification, severity stratification, relation to cytokine elaboration and outcome prediction in posttrauma critical illness. J Trauma. 1996 Oct;41(4):581-98. doi: 10.1097/00005373-199610000-00001. PMID 8858015
- [Background] Convertino VA, Howard JT, Hinojosa-Laborde C, Cardin S, Batchelder P, Mulligan J, Grudic GZ, Moulton SL, MacLeod DB. Individual-Specific, Beat-to-beat Trending of Significant Human Blood Loss: The Compensatory Reserve. Shock. 2015 Aug;44 Suppl 1:27-32. doi: 10.1097/SHK.0000000000000323. PMID 25565640
- [Background] Nadler R, Convertino VA, Gendler S, Lending G, Lipsky AM, Cardin S, Lowenthal A, Glassberg E. The value of noninvasive measurement of the compensatory reserve index in monitoring and triage of patients experiencing minimal blood loss. Shock. 2014 Aug;42(2):93-8. doi: 10.1097/SHK.0000000000000178. PMID 24667628